CLINICAL TRIAL: NCT00504959
Title: A Phase IV, Long-term, Open-label, Multicenter Extension Study to Evaluate the Safety and Tolerability of Ranibizumab in Patients With Subfoveal Choroidal Neovascularization (CNV) Secondary to Age-related Macular Degeneration (AMD)
Brief Title: Safety and Tolerability of Ranibizumab in Patients With Subfoveal Choroidal Neovascularization Secondary to Age-related Macular Degeneration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002A2402
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Subfoveal Choroidal Neovascularization (CNV); Secondary to Age-related Macular Degeneration (AMD)
Keywords: Age-related macular degeneration (AMD),; choroidal neovascularization (CNV),; vascular endothelial growth factor (VEGF)
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Ranibizumab

ARMS (1):
- 1 (Experimental): ranibizumab
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab
  Other Names: rhuFab V2, Lucentis

SUMMARY:
This extension study will investigate the long-term safety and tolerability of multiple intravitreal injections of ranibizumab administered to patients with subfoveal choroidal neovascularization secondary to age-related macular degeneration who have been previously treated in either of the two ongoing ranibizumab studies CRFB002A2302 (EXCITE) or CRFB002A2303 (SUSTAIN

ELIGIBILITY:
Inclusion Criteria:

* Completion of 12-month treatment period of study CRFB002A2302 (EXCITE) or CRFB002A2303

Exclusion Criteria:

* Concurrent participation in another clinical trial, i.e. use of other investigational drugs

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety assessed by incidence and severity of treatment emergent ocular and non-ocular adverse events over 24 month study period with ranibizumab monthly prn (0.5mg/0.05ml)

SECONDARY OUTCOMES:
Efficacy assessed by mean change in BCVA from Baseline at M 6, 12, 18, and 24. Number of injections with ranibizumab. Safety assessed by AEs and SAEs leading to premature discont. of study drug, vital signs, and ophthalmic exams.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Board of Hacettepe University , Ankara, turkey
Locations (36):
- Novartis Investigational Site, Melbourne, Australia
- Belgium (3):
  - Novartis Investigative Site, Laken
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Germany (13):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Siegburg
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Würzburg
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Israel (3):
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Tel Litwinsky
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Nijmegen
- Portugal (2):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Porto
- Spain (5):
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Valencia
- Novartis Investigative SIte, Ankara, Turkey (Türkiye)
- United Kingdom (4):
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, West Midlands
  - Novartis Investigative Site, Wolverhampton

REFERENCES:
- [Derived] Silva R, Axer-Siegel R, Eldem B, Guymer R, Kirchhof B, Papp A, Seres A, Gekkieva M, Nieweg A, Pilz S; SECURE Study Group. The SECURE study: long-term safety of ranibizumab 0.5 mg in neovascular age-related macular degeneration. Ophthalmology. 2013 Jan;120(1):130-9. doi: 10.1016/j.ophtha.2012.07.026. Epub 2012 Sep 25. PMID 23021093